#### **CONSENT FOR RESEARCH**

The Pennsylvania State University

| Title of Project: Testing a Smartphone Intervention for Anxiety and Learning |
|---|
| Principal Investigator: Lucas S. LaFreniere, M.S. |
| Address: 378 Moore Building, The Pennsylvania State University, University Park, PA 16801 |
| Advisor: Michelle Newman, Ph.D. |
| Subject's Printed Name: |

We are asking you to be in a research study. This form gives you information about the research.

Whether or not you take part is up to you. You can choose not to take part. You can agree to take part and later change your mind. Your decision will not be held against you.

Please ask questions about anything that is unclear to you and take your time to make your choice.

### 1. Why is this research study being done?

We are asking you to be in this research because of your scores on anxiety surveys in the subject pool screening, which were either high or low. This research is being done to find out if a smartphone-assisted intervention undertaken in participant's daily lives can reduce worry and anxiety, increase positive feelings and well-being, and improve participants' ability to learn by feedback. Approximately 250 people will take part in this research study here at Penn State.

### 2. What will happen in this research study?

In this study you will be asked to do a variety of tasks in this lab and in daily life by smartphone. The study will have two parts—a first part across six days that all participants will complete for partial credit and a second part for full credit across four days for participants who sufficiently completed the tasks in the first part. If participants engage in the first part sufficiently, they will be invited to the second part.

First, you will be asked to undergo a session of questionnaires, a computerized task, and an intervention training for one hour and 30 minutes. In this session you will be asked to complete a series of questionnaires on a computer asking about your levels of worry, anxiety, positive feelings, responses to positive feelings, and thinking tendencies. In all the questionnaires in this study, you are free to skip any questions that you would prefer not to answer. Afterward, you will be asked to undergo a task in which you will repeatedly attempt to choose the correct symbol from a pair of symbols. After each choice, you will receive feedback via the appearance or absence of a happy face image. After repeated trials of this task you will complete a few questions about the experiment. Lastly, you will be asked to undergo training for using a smartphone-assisted intervention. In this training you will download and be instructed in the use of two free smartphone apps (PACO and Quip). You will then be guided through exercises to practice remembering positive memories, attending to and holding onto positive feelings, brainstorming and scheduling enjoyable activities, and reflecting on what you are looking forward to in your day.

You will then be asked to use a smartphone-assisted intervention over the following 4 days. This intervention has been designed to increase enjoyable thinking about the past, present, and future and increase paying full attention to, planning, and participating in enjoyable experiences. It will involve five aspects: Planning and engaging in enjoyable activities, savoring positive memories, thinking and writing briefly about what went well in your day, paying attention to the good aspects of the present moment, and imagining your best possible future. These aspects will be guided by randomly-timed notifications and surveys between 9AM and 11PM on your smartphone through the apps previously mentioned.

On the fifth day of the study you will receive a phone call that will ask several questions. This call will determine whether you can continue on to the second part of the study and receive full credit. You must answer this call and have completed a high number of prompts and study activities to continue to part two. If you have completed enough prompts, you will be invited to complete three more days of the intervention activities. That same day (the fifth day) you will be asked to complete a short series of questionnaires online in any location you choose. On the eighth day of the study you will be asked to return to the laboratory for half an hour and complete another series of questionnaires and a similar computerized learning task. Lastly, thirty days after your first session you will be asked by email to complete another series of questionnaires for twenty minutes in any location you would prefer.

### 3. What are the risks and possible discomforts from being in this research study?

This study is of minimal risk to those participating, yet participants may experience a few foreseeable discomforts. There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your electronic data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed. In addition, thinking about and reporting about worries and anxiety and changing your thoughts may lead to some unpleasant emotions. If any feelings or thoughts arise that you would like to address with a mental health professional, feel free to call the Penn State Psychological Clinic at **814-865-2191** or Penn State Counseling and Psychological Services (CAPS) at **814-863-0395** to set up an appointment.

# 4. What are the possible benefits from being in this research study? 4a. What are the possible benefits to you?

The potential benefits to you are a possible decrease in worrying, anxiety, and depressive feelings, a possible increase in how often, for how long, and how intensely you experience positive feelings, and a possible improvement in your basic learning ability through the use of the intervention.

### 4b. What are the possible benefits to others?

The potential benefits to society include a better understanding of the influence of this intervention, positive emotions in general, and pleasurable activity scheduling on anxiety and depression. This information may help psychologists determine how to better treat worry and anxiety.

#### 5. What other options are available instead of being in this research study?

You may decide not to participate in this research. Since the Penn State Psychology subject pool will be used to recruit participants, you will receive course credit for participating as specified in your instructor's syllabus. Alternative means for earning this credit are available as specified in the syllabus.

### 6. How long will you take part in this research study?

If you agree to take part and complete study tasks sufficient by the fifth day, it will take you about a total of **6 hours** spread across 30 days to complete this study. You will be asked to return to the research site two times, once for a one and a half hour session and once for a 30-minute session. You will also undertake the intervention for approximately 28 minutes total each day for seven days (approximately 3 hours, 15 minutes). Lastly, you will spend approximately 35 minutes taking questionnaires online in any location you choose. Those who do not sufficiently complete study tasks by the fifth day and do not proceed will have a total participation time of approximately 3 hours and 30 minutes.

# 7. How will your privacy and confidentiality be protected if you decide to take part in this research study?

Efforts will be made to limit the use and sharing of your personal research information to people who have a need to review this information.

- A list that matches your name with your code number will be kept in a locked file or password protected file in Moore Building laboratory rooms or study computers.
- Your research records will be labeled with your code number and will be kept in a locked location and password protected electronic files in Moore Building laboratory rooms.

In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

We will do our best to keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people may find out about your participation in this research study. For example, the following groups may check and copy records about this research.

- The Office for Human Research Protections in the U. S. Department of Health & Human Services
- The Institutional Review Board (a committee that reviews and approves research studies) and
- The Office for Research Protections.

Some of these records could contain information that personally identifies you. Reasonable efforts will be made to keep the personal information in your research record private. However, absolute confidentiality cannot be guaranteed.

## 8. Will you be paid or receive credit to take part in this research study?

<u>Subject Pool Participants ONLY receiving credit:</u> You will receive course credit for participating as specified in the syllabus provided by your instructor. You may receive up to 6 subject pool credits. You will receive 3.5 subject pool credit hours for completion of the first part of the study (prior to the fifth day of intervention use). If you sufficiently complete study tasks up to the fifth day compliance check, you will be invited to finish the second part of the study and receive an additional 2.5 subject pool credit hours. Alternative means for earning this course credit are available as specified in the syllabus.

<u>Subject Pool Participants receiving credit plus monetary compensation</u>: For participating, you will first receive the remaining course credit hours you need to reach your required 6. This is the number of credits you need to reach 6 total course credits across all subject pool studies in which you have participated. Please enter that the number of credits you still need to reach 6 here \_\_\_\_\_\_. After

receiving these credit hours, you will receive up to \$5.00 for each additional hour you spend in the study. The more study responses and tasks you complete, the more money you will make. The amount you will receive will be the percentage of study tasks and responses to smartphone prompts multiplied by \$5.00 for each remaining hour of participation. In other words, you will first receive your remaining needed credit hours. You will then receive a percentage of \$5.00 for each remaining hour of participation, which is the percentage of study tasks and responses you complete. Here is an equation that will be used to calculate your final compensation amount: [credit hours + (% task completion x (\$5.00 x your remaining hours of participation))].

You cannot start receiving money until all of your needed credit hours are completed first (for a total of at least 6 hours). You will receive 3.5 subject pool credit hours for completion of the first part of the study (prior to the fifth day of intervention use). If you sufficiently complete study tasks up to the fifth day compliance check, you will be invited to finish the second part of the study and receive an additional 2.5 subject pool credit hours (up to your total of 6) OR your task completion percentage multiplied by \$5.00 for each remaining hour.

As an example, if you only needed 2 more credit hours to reach your total of 6, then completed 90% of tasks/prompts in study's last 4 hours, you would get 2 credit hours plus  $.90 \times (5 \times 4 \text{ hours}) = $18.00$ 

Alternative means for earning this course credit are available as specified in the syllabus.

## Those participating ONLY for money or subject pool participants who have completed all 6 credits:

You will be paid up to \$30.00 for your participation in this study. The more study tasks and responses you complete, the more money you will receive. You will receive \$30.00 times the the percentage of study tasks and responses to smartphone prompts that you complete. In other words, you will receive \$5.00 per hour of participation multiplied by the percentage of study tasks/prompts you complete. The maximum is \$30.00 ( $$5 \times 6$  hours). You can receive up to \$17.50 for 100% completion of the first part of the study (prior to the fifth day of intervention use). If you sufficiently complete study tasks up to the fifth day compliance check, you will be invited to finish the second part of the study. In this second part of the study, you will have to opportunity to receive an additional \$12.50 with 100% completion.

As an example, if you complete 93% of study tasks and complete all 6 hours of participation, you will receive  $.93 \times (\$5.00 \times 6 \text{ hrs}) = \$27.90$ . The more prompts you complete, the more money you make.

### 9. What are your rights if you take part in this research study?

Taking part in this research study is voluntary.

- You do not have to be in this research.
- If you choose to be in this research, you have the right to stop at any time.
- If you decide not to be in this research or if you decide to stop at a later date, there will be no penalty or loss of benefits to which you are entitled.

If any new information arises during the study that may affect your health, welfare, or your decision to continue participating in this research, you will be provided with that information.

### 10. If you have questions or concerns about this research study, whom should you call?

Please call the head of the study (principal investigator), Lucas LaFreniere at (906) 361-6958 if you:

- Have questions, complaints, or concerns about the research.
- Believe you may have been harmed by being in the research study.

You may also contact the Office for Research Protections at (814) 865-1775, ORProtections@psu.edu if you:

- Have questions regarding your rights as a person in a research study.
- Have concerns or general questions about the research.
- You may also call this number if you cannot reach the research team or wish to talk to someone else about any concerns related to the research.

# INFORMED CONSENT TO TAKE PART IN RESEARCH

## **Signature of Person Obtaining Informed Consent**

| Your signature below means that you representative and have answered a | • | |
|---|---|---|
| Signature of person who explained this | | Printed Name |
| Signature of Person Giving Informed | | esearch and obtain informed consent.) |
| - | with an investigator, form, and may have questions you may have have received this informates the stions have been answer | |
| Signature of Subject | | |
| By signing this consent form, you indicallow your information to be used and | • | noose to be in this research and agree to ve. |
| Signature of Subject | <br>Date | Printed Name |